CLINICAL TRIAL: NCT01040702
Title: The Effect of Methylphenidate on Decision-making Ability of ADHD Adults
Brief Title: The Effect of Methylphenidate on Decision-making Ability of Attention Deficit Hyperactivity Disorder (ADHD) Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Ziv Carmel,MD, Shalvata MHC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SH-40107
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2009-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Sweetening Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ADHD -MPH (Experimental): adults with ADHD diagnosis who receive a single dose of Methylphenidate
  Interventions: Drug: methylphenidate
- ADHD-placebo (Placebo Comparator): adults with ADHD diagnosis who received placebo
  Interventions: Dietary Supplement: sweetener pill
- non-ADHD-MPH (Experimental): healthy adults who received a single dose of Methylphenidate
  Interventions: Drug: methylphenidate
- non-ADHD-placebo (Placebo Comparator): healthy adults who received placebo
  Interventions: Dietary Supplement: sweetener pill

INTERVENTIONS:
Drug: methylphenidate — a single doses of 10-20 mg in each one of two visits
  Other Names: Ritalin
  Arms: ADHD -MPH; non-ADHD-MPH
Dietary Supplement: sweetener pill — a capsule containing a sweetener pill
  Other Names: sukrazit
  Arms: ADHD-placebo; non-ADHD-placebo

SUMMARY:
The aim of the study is to assess the effect of Methylphenidate on cognitive performance and decision-making ability of ADHD adults, and to compare this effect to the effect on healthy control adults.

DETAILED DESCRIPTION:
Two matched groups of adults - with and without ADHD diagnosis - will perform a battery of computerized tasks assessing sustained attention,working-memory,non-verbal IQ,and decision-making ability. In each group,half of the participants will perform the tasks after receiving a capsule containing methylphenidate (MPH), and the other half will perform the tasks after receiving placebo. Task performance measures will then be compared in order to assess the effect of MPH on these domains.

ELIGIBILITY:
Inclusion Criteria:

* adults in the age of 21-50

Exclusion Criteria:

* pregnant or nursing women.
* people who suffer from a psychiatric disorder other than ADHD which could account for their inattention symptoms better than ADHD.
* people who lack judgment or are unable to communicate with the experimenters.
* people who are incapable of performing the computerized tasks due to sensory or motor disabilities.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
score in decision-making task 1 | by the end of the task

SECONDARY OUTCOMES:
working memory task score | by the end of the task

CONTACTS AND LOCATIONS:
Overall Officials: Ziv Carmel, MD, Principal Investigator — MD
Locations (1):
- cognitive laboratory,Shalvata MHC, Hod HaSharon, Israel